CLINICAL TRIAL: NCT02941939
Title: Effects of High-Intensity Interval Training (HIT) While in a Hyperoxic-Hyperbaric Environment on Exercise Performance (HITOP Study)
Brief Title: Effects of High-Intensity Interval Training (HIT) While in a Hyperoxic-Hyperbaric Environment on Exercise Performance
Acronym: HITOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1050188
Record Dates: First submitted 2016-10-10; First posted 2016-10-21 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Exercise Performance
Keywords: high intensity interval training; hyperbaric oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ambient pressure arm (Active Comparator): High intensity training will be completed while the subjects are breathing normal air.
  Interventions: Other: Ambient pressure
- Hyperoxic-hyperbaric arm (Experimental): The high intensity training program will be carried out in a hyperbaric chamber.
  Interventions: Other: Hyperbaric chamber

INTERVENTIONS:
Other: Hyperbaric chamber
  Arms: Hyperoxic-hyperbaric arm
Other: Ambient pressure
  Arms: Ambient pressure arm

SUMMARY:
Hyperbaric oxygen has previously been tested as a possible means for pre-conditioning to enhance exercise performance. This study is designed to examine the effects of exercising in a hyperbaric chamber for improving fitness when combined with high-intensity training.

DETAILED DESCRIPTION:
The purpose of this research study is to determine the incremental benefit of high intensity interval training (HIT) in a hyperbaric-hyperoxic environment with HIT alone in healthy subjects and to compare the effect of HIT at an intermediate altitude (SLC, UT; altitude 1420 m) with that performed at sea-level (Durham, NC) in healthy subjects. While VO2 max is determined by the functional interdependence of the respiratory, cardiovascular and muscular systems, ultimately VO2 max is determined by mitochondrial oxidative capacity. Exercise training increases mitochondrial capacity. There is evidence that high intensity interval training (HIT) programs are effective at increasing exercise capacity. Furthermore, there is evidence that training while in a hyperbaric-hyperoxic environment may potentiate the HIT training effect through its effects on mitochondrial oxidative capacity, but this has not been scientifically tested. Our hypothesis is that high intensity interval training (HIT) in a hyperoxichyperbaric environment performed six-times over a two-week period will increase exercise performance compared with HIT performed in ambient conditions in healthy subjects. The primary outcome studied will be the effect of high-volume interval training in a hyperbaric-hyperoxic on VO2max.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals, ages 18-40 years that are sedentary or recreationally active but not involved in any structured endurance training will be eligible for the study. This level of activity will be defined as performing mild-moderate aerobic exercise 0-3 times per week.
* VO2 max within normal limits (defined as 84-120% predicted using Wasserman reference equations48).
* Spirometry within predicted limits.

Exclusion Criteria:

* Subjects unable to complete a satisfactory VO2 max test
* Individuals with chronic cardiovascular disease such as hypertension, valve disease, coronary artery disease, cardiac conduction abnormalities, etc.
* History of pneumothorax or chronic lung disease such as asthma, COPD, bronchiectasis
* Active Smokers
* Pregnant women
* Persons unable to read or understand English, not in full mental capacity or suffer from blindness.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2016-04-14 (Actual); Primary Completion 2017-04-08 (Actual); Study Completion 2017-06-08 (Actual)

PRIMARY OUTCOMES:
Change in maximum VO2 at 2 weeks compared to baseline | 2 weeks
  Comparison of post-training VO2 results with baseline in the two HIT groups (performed at ambient conditions in Salt Lake City, UT and hyperbarichyperoxic conditions); the results of HIT at Salt Lake City, UT altitude will be compared with those performed at sea-level altitude in Durham, NC.

SECONDARY OUTCOMES:
Change in VO2 measured at anaerobic threshold (in mL O2/kg/min) at 2 weeks compared to baseline | 2 weeks
  Difference post-training minus pre-training
ΔVO2/ΔWR (in mL O2/kg/min/Watt; a measure of exercise efficiency) | 2 weeks
  Difference post-training minus pre-training
Change in peak work rate (in Watts) at 2 weeks compared to baseline | 2 weeks
  Difference post-training minus pre-training
Change in heart rate response to exercise at 2 weeks compared with baseline | 2 weeks
  Difference post-training minus pre-training
Change in level of perceived exertion at 2 weeks compared with baseline | 2 weeks
  Difference post-training minus pre-training
Change in Borg dyspnea score at 2 weeks compared with baseline | 2 weeks
  Difference post-training minus pre-training

CONTACTS AND LOCATIONS:
Overall Officials: Matt Hegewald, MD, Principal Investigator — Intermountain Health Care, Inc.
Locations (1):
- Intermountain Medical Center, Murray, Utah, United States

IPD SHARING:
Plan to Share IPD: No